CLINICAL TRIAL: NCT01441817
Title: Non--operative Treatment of the Medial Malleolus in bi- and Trimalleolar Ankle Fractures. A Randomized Controlled Trial
Brief Title: Non--operative Treatment of the Medial Malleolus in bi- and Trimalleolar Ankle Fractures
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Oslo University Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 224-01077(REK); REK (Other: 224-01077)
Record Dates: First submitted 2011-09-15; First posted 2011-09-28 (Estimated); Last update posted 2011-09-28 (Estimated); Status verified 2011-09

CONDITIONS: Ankle Malleolus Fracture Bimalleolar; Fracture of Medial Malleolus; Fracture of Ankle
MeSH Terms: conditions — Ankle Fractures | interventions — Fracture Fixation, Internal

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Surgery (Other)
  Interventions: Procedure: Internal fixation

INTERVENTIONS:
Procedure: Internal fixation — Internal fixation of the medial malleolus following open reduction and internal fixation of the lateral and, if required, posterior malleolus.

SUMMARY:
The purpose of this study was to determine if internal fixation of the medial malleolus is necessary following open reduction and internal fixation of the lateral and, if required, the posterior malleolus treating displaced bi-or trimalleolar ankle fractures.

ELIGIBILITY:
Inclusion Criteria:

* Patients with Orthopaedic Trauma Association (OTA) type 44 fractures (B2-3 and C2-3).

Exclusion Criteria:

* Patients with OTA type 43 distal tibia fractures.
* Patients with soft tissue injuries involving the medial malleolus.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2002-05; Primary Completion 2008-08 (Actual); Study Completion 2008-08 (Actual)

PRIMARY OUTCOMES:
American Orthopaedic Foot and Ankle Society ankle hind foot score (AOFAS) | Average of 42 months
The Olerud Molander Ankle score (OMAS) | Average of 42 months

SECONDARY OUTCOMES:
Posttraumatic osteoarthritis (OA) according to the criteria of Magnusson (stage I-IV) | Average of 42 months
VAS score | Average of 42 months
  Pain evaluated at rest, in the morning, in the evening and during the night.

CONTACTS AND LOCATIONS:
Locations (1):
- Oslo University Hospital, Oslo, Norway